CLINICAL TRIAL: NCT00225797
Title: An Open-Label Titration Followed by a Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Tolerability, and Safety of Oxymorphone Extended Release Tablets in Opioid-Naïve Patients With Chronic Low Back Pain
Brief Title: Efficacy and Safety of Oxmorphone Extended Release in Chronic Non-malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director Clinical R&D
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3202-031
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain
Keywords: chronic pain; lower back; opioid; efficacy; safety
MeSH Terms: conditions — Chronic Pain

INTERVENTIONS:
Drug: Oxymorphone Extended Release

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy and safety of oxymorphone extended release in non-cancer patients with chronic low back pain.

DETAILED DESCRIPTION:
Patients with low back pain who are sub-optimally responsive to their current analgesic treatment begin open-label treatment with oxymorphone extended release (ER). During the Open-Label Titration Period, patients will receive daily oxymorphone ER by mouth (PO) q12h. The investigator will initiate the Open-Label Titration Period using study drug at a dose of 5 mg PO q12h for 2 days; thereafter, patients will continue receiving 5 mg q12h or be titrated at increments of 5-10 mg q12h every 3-7 days until stabilization is achieved. The goal of the Open-Label Titration Period is to determine for each patient a fixed dose of study medication that is tolerated and achieves adequate analgesia. Stabilized patients will be randomiozed to either continue with current dose of oxymorphone ER or receive placebo for a total duration of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older
* opioid naïve
* Have an initial pain intensity score of at least 50 mm VAS
* In good health as determined by the investigator on the basis of medical history and physical examination
* Have moderate to severe chronic non-neuropathic LBP that has been present daily for at least several hours per day for a minimum of three months prior to the Screening
* Any adjunct therapy for back pain such as physical therapy, biofeedback therapy, acupuncture therapy or herbal remedies, based on the patient's current status should remain unchanged during the period of participation of the patient
* Written informed consent

Exclusion Criteria:

* Pregnant and/or lactating
* Radiculopathy, fibromyalgia, reflex sympathetic dystrophy or causalgia (complex regional pain syndrome), acute spinal cord compression, cauda equina compression, acute nerve root compression, severe lower extremity weakness or numbness, bowel or bladder dysfunction secondary to cauda equina compression, diabetic amyotrophy, meningitis, discitis, or back pain due to secondary infection or tumor
* Cannot or will not agree to stop local regional pain treatments during the study (nerve/plexus blocks or ablation, neurosurgical procedures for pain control, or inhalation analgesia). The patient must not have a nerve/plexus block within 4 weeks of screening
* Intend to alter physical therapy regimen during the study.
* Surgical procedures directed towards the source of back pain within 6 months of screening
* Pain which is secondary to confirmed or suspected neoplasm
* Dysphagia or difficulty swallowing tablets or capsules, or an inability to take oral medication
* Significant prior history of substance abuse or alcohol abuse
* Use of any investigational medication within 30 days prior to the first dose of study medication
* Previous exposure to oxymorphone
* History of clinically significant intolerance to oxymorphone or a known hypersensitivity to opioid analgesics
* History of seizure
* Ileostomy or colostomy
* Use of MAO inhibitor within 14 days prior to the start of study medication
* Other clinically significant conditions as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2004-11; Study Completion 2005-07

PRIMARY OUTCOMES:
Change in pain intensity from baseline (pre-randomization) to last assessment.

SECONDARY OUTCOMES:
Time to early discontinuation due to lack of efficacy
Patient's Global Assessment of Pain Medication
Physician's Global Assessment of Pain Medication
Safety as measured by AEs

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Southern Drug Research, Hueytown, Alabama
  - Phoenix Center for Clinical Research, Phoenix, Arizona
  - Express Care Clinical Research, Colorado Springs, Colorado
  - New England Research, Bridgeport, Connecticut
  - Glasgow Family Practice, Newark, Delaware
  - Radiant Research, Daytona Beach, Florida
  - University Clinical Research, DeLand, Florida
  - LCFP Inc, Fort Myers, Florida
  - Century Clinical Research, Holly Hill, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Radiant Research, Pinellas Park, Florida
  - Park Place Therapeutic Center, Plantation, Florida
  - ICSL Clinical Studies, St. Petersburg, Florida
  - Comprehensive Neurology Specialists, Atlanta, Georgia
  - Comprehensive Neuroscience, Atlanta, Georgia
  - Pain Specialists of Greater Chicago, Burr Ridge, Illinois
  - Mid-America Physiatrists, Overland Park, Kansas
  - Research Medical Center, Kansas City, Missouri
  - Radiant Research, St Louis, Missouri
  - Piedmont Anesthesia, Winston-Salem, North Carolina
  - Keystone Clinical Solutions, Altoona, Pennsylvania
  - Perkiomen Valley Family Practice, Collegeville, Pennsylvania
  - Feasterville Family Health Center, Feasterville, Pennsylvania
  - Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Paragon Clinical Research, Cranston, Rhode Island
  - Radiant Research, Greer, South Carolina
  - Waccamaw Pain Management, Murrells Inlet, South Carolina
  - KRK Medical Research, Richardson, Texas
  - Intermountain Clinical Research, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Peniston JH, Hu X, Potts SL, Wieman MS, Turk DC. Tolerability of concomitant use of selective serotonin reuptake inhibitors or serotonin-norepinephrine reuptake inhibitors and oxymorphone extended release. Postgrad Med. 2012 Mar;124(2):114-22. doi: 10.3810/pgm.2012.03.2542. PMID 22437221
- [Derived] Peniston JH, Xiang Q, Gould EM. Factors affecting acceptability of titrated oxymorphone extended release in chronic low back pain - an individual patient analysis. Curr Med Res Opin. 2010 Aug;26(8):1861-71. doi: 10.1185/03007995.2010.490457. PMID 20521870
- [Derived] Katz N, Rauck R, Ahdieh H, Ma T, Gerritsen van der Hoop R, Kerwin R, Podolsky G. A 12-week, randomized, placebo-controlled trial assessing the safety and efficacy of oxymorphone extended release for opioid-naive patients with chronic low back pain. Curr Med Res Opin. 2007 Jan;23(1):117-28. doi: 10.1185/030079906x162692. PMID 17257473